CLINICAL TRIAL: NCT01094769
Title: Sympathetic Nervous System Inhibition for the Treatment of Diabetic Nephropathy
Brief Title: Sympathetic Nervous System Inhibition for the Treatment of Diabetic Kidney Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 101/10; 58667 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2010-03-26; First posted 2010-03-29 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — moxonidine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxonidine (Experimental)
  Interventions: Drug: Moxonidine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxonidine — Patients will receive moxonidine treatment for 12 weeks, at a dose of 0.4mg/d for the first 6 weeks of treatment followed by up-titration of the dose to 0.6 mg/d for the final 6 weeks.
  Other Names: Physiotens
  Arms: Moxonidine
Drug: Placebo — lactose capsule taken once daily
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether moxonidine is effective in reducing urine albumin levels in patients with diabetic kidney disease.

DETAILED DESCRIPTION:
This study will investigate the effect of moxonidine in lowering urine albumin excretion and limiting further damage to the kidneys in patients with diabetic nephropathy. Reducing urine albumin excretion in type 2 diabetic patients is an indicator of successful treatment. Previous studies have shown that drugs that work in a similar fashion to moxonidine (intervene with the sympathetic nervous system)have been very effective in reducing the amount of albumin in the urine and are associated with long term renal and cardiovascular protection.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-75 years
* diabetic nephropathy as defined by the mean of three consecutive early morning urinary albumin-creatinine ratios (UACR) of >300mg per gram, or > 200mg per gram in patients receiving therapy targeted at blockade of the RAS

Exclusion Criteria:

* non-diabetic kidney disease
* UACR of more than 3500mg per gram, an estimated glomerular filtration rate of less than 30ml/min/1.73m2.
* chronic urinary tract infection.
* severe hypertension
* heart failure New York Heart Association (NYHA) class II-IV
* major cardiovascular disease within the previous 6 months
* left ventricular ejection fraction <55%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-04; Primary Completion 2020-01 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Urine albumin/creatinine ratio (UACR) | 12 weeks
  The primary outcome measure is the difference in the change of UACR between active treatment and placebo from baseline to week 12 of treatment.

SECONDARY OUTCOMES:
muscle sympathetic nerve activity (MSNA) | 12 weeks
  Secondary outcome measure is the difference between active and placebo treatment in the change from baseline to week 12 of treatment in muscle sympathetic nerve activity

CONTACTS AND LOCATIONS:
Overall Officials: Markus P Schlaich, MD, Principal Investigator — Baker Heart and Diabetes Institute; Gavin W Lambert, BSc PhD, Principal Investigator — Baker Heart and Diabetes Institute
Locations (1):
- Alfred & Baker Medical Unit, Melbourne, Victoria, Australia